CLINICAL TRIAL: NCT02028949
Title: LIDA-B: Treatment of Cirrhosis-related Hepatocellular Carcinoma With the Intrahepatic Arterial Injection of an Emulsion of Lipiodol and Idarubicin (Zavedos®): Phase I Study
Brief Title: Treatment of Cirrhosis-related Hepatocellular Carcinoma With the Intrahepatic Arterial Injection of an Emulsion of Lipiodol and Idarubicin (Zavedos®): Phase I Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None
Other Study IDs: GUIU APJ 2012
Record Dates: First submitted 2013-12-18; First posted 2014-01-07 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Unresectable Non-metastatic Hepatocellular Carcinoma; Child A/B7 Cirrhosis
MeSH Terms: interventions — Idarubicin; Blood Specimen Collection

ARMS (1):
- Chemo-lipiodol (Experimental)
  Interventions: Drug: Zavedos®; Other: Blood samples

INTERVENTIONS:
Drug: Zavedos®
Other: Blood samples

SUMMARY:
Unresectable, non-metastatic cirrhosis-related hepatocellular carcinoma (HCC) has a poor prognosis as there are no recommended curative treatments. Chemoembolisation is the most widely used treatment in these patients, but this technique can prove to be toxic. intrahepatic arterial chemotherapy with lipiodol and idarubicin could be an effective therapeutic approach, without deteriorating liver function.

The rationale for this treatment can be resumed as follows:

* HCC are vascularised via the hepatic artery system
* The IHA perfusion of anthracyclines leads to high elimination via the liver with low systemic concentrations
* The absence of embolisation reduces toxicity
* the toxiciity profile of idarubicin is well known and the drug is widely used for the IV treatment of leukemia
* idarubicin is the most cytotoxic drug for tumor cell lines.
* The in vitro cytotoxicity of idarubicin is 100% at low concentrations
* Lipiodol can stay in contact with tumor tissue for several weeks after injection and act as a vector for the drug
* The idarubicin-lipiodol is more stable than lipidol emulsions usually given by intraarterial injection
* The emulsion is more stable with idarubicin than with other anticancer molecules
* Sequential inclusion in accordance with the "continual reassessment method" makes it possible to increase inclusions at a target toxicity level while reducing inclusions at doses that are too low or too toxic The aim of the treatment is to improve survival.

ELIGIBILITY:
Inclusion criteria:

Histologically-proven hepatocellular carcinoma or carcinoma meeting validated non-invasive criteria (EASL, AASLD)

* Child-Pugh A OR B7 cirrhosis
* General health status WHO 0.1
* Platelets > 50 000/mm3, Polynuclear neutrophils > 1000/mm3
* Creatininemia < 1.5 times upper limit of normal
* LVEF by MUGA scan or US > 50 %
* Age > 18 years
* Signed informed consent
* For women child-bearing age, an effective means of contraception

Exclusion criteria:

Patients who can benefit from curative treatment (surgical resection, liver transplant or treatment via percutaneous destruction)

* Non-cirrhotic liver
* Cirrhosis Child B8 or B9 or C
* Extrahepatic metastases (pulmonary micronodules < 7mm are not considered a contra-indication)
* Digestive hemorrhage within the previous month
* Patient on anticoagulants
* Pregnant women
* Uncontrolled infection
* Hypersensitivity to anthracyclines
* Hypersensitivity to iodine contrast agents
* Patient under guardianship or ward of court
* Patients who have already received the recommended cumulative dose of anthracycline (93 mg/m2 for idarubicin, 140 mg/m2 for mitoxantrone, 550 mg/m2 for doxorubicin, 600 mg/m2 for daunorubicin, 900 mg/m2 for epirubicin)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11-22 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-02-05 (Actual)

PRIMARY OUTCOMES:
tolerance: toxicity will be evaluated according to the NCI CTC AE version 4.03 scale to determine the limiting dose | 7 weeks after the 2 injections

SECONDARY OUTCOMES:
Study the pharmacokinetics of idarubicin in this delivery method | 24 months
Evaluate overall survival | 24 months
Evaluate progression-free survival | 24 months
Evaluate time to progression | 24 months
Evaluate the rate of objective response | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France

REFERENCES:
- [Result] Guiu B, Jouve JL, Schmitt A, Minello A, Bonnetain F, Cassinotto C, Piron L, Cercueil JP, Loffroy R, Latournerie M, Wendremaire M, Lepage C, Boulin M. Intra-arterial idarubicin_lipiodol without embolisation in hepatocellular carcinoma: The LIDA-B phase I trial. J Hepatol. 2018 Jun;68(6):1163-1171. doi: 10.1016/j.jhep.2018.01.022. Epub 2018 Feb 8. PMID 29427728